CLINICAL TRIAL: NCT05871879
Title: Association Between Frailty and Postoperative Adverse Outcomes in Patients Undergoing Urological Surgery
Status: Completed | Type: Observational
Sponsor: Taipei Medical University Hospital (Other)
Responsible Party: Principal Investigator, Chao-Shun Lin, Attending physician of anesthesiology, clinical professor, Taipei Medical University Hospital
Other Study IDs: 202305015
Record Dates: First submitted 2023-05-15; First posted 2023-05-23 (Actual); Last update posted 2023-05-23 (Actual); Status verified 2023-05

CONDITIONS: Frailty; Postoperative Complications
Keywords: Frailty; Postoperative Complications; Urologic Surgery
MeSH Terms: conditions — Frailty; Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- All adult patients who underwent urologic procedures: The included procedures included all urologic oncology surgeries, suburethral sling placement, laparoscopic pyeloplasty, transurethral resection of the prostate, transurethral resection of the bladder tumor, ureteroscopy, hydrocelectomy, orchiectomy, spermatocelectomy, epididymectomy, and varicocelectomy.
  Interventions: Diagnostic Test: The 5-item modified frailty index

INTERVENTIONS:
Diagnostic Test: The 5-item modified frailty index — The mFI-5 contains five items, including hypertension, diabetes, congestive heart failure (CHF), chronic obstructive lung disease (COPD), and physical function status, with each item attributing 1 point. Patients with an mFI-5 score greater than or equal to 2 were considered frail, while those with an mFI-5 score of 0 or 1 were considered nonfrail.
  Other Names: mFI-5

SUMMARY:
Frailty is a clinical condition associated with aging that is characterized by a decline in physiological capacity involving multiple organ systems. Previous research has established a strong correlation between frailty and increased mortality and morbidity risk after surgery. The 5-item modified frailty index (mFI-5) is a recent tool used to assess frailty. The aim of the present study was to use the mFI-5 to identify frailty and its association with postoperative adverse outcomes, including mortality and morbidity, among patients who underwent urologic procedures.

DETAILED DESCRIPTION:
Frailty is a clinical condition that often develops with age and is characterized by a decline in physiological capacity and dysfunction across multiple organ systems. This decline results in reduced physical reserve and an increased vulnerability to acute stressors, such as surgical interventions. The prevalence of frailty varies based on the definition used, with 15% of the nonnursing home population in the US experiencing frailty and 45% experiencing prefrailty. Frailty is more common in individuals with certain comorbidities, such as HIV infection, chronic obstructive pulmonary disease, and end-stage renal disease, and it is more prevalent with increasing age.

Previous studies have established a link between urologic issues and frailty. In fact, more than 40% of patients with lower urologic symptoms exhibit frailty-related features such as sarcopenia, dysmotility, multimorbidity, and a heightened risk of malnutrition. Additionally, common geriatric ailments, such as benign prostate hypertrophy, dementia, spinal disc herniation, and cerebral infarction, are also associated with neurogenic bladder and other voiding difficulties. Consequently, surgical intervention is often necessary for these populations. However, even minimally invasive procedures may be risky due to the vulnerability of frail individuals. Prior studies have shown a strong correlation between frailty and the likelihood of postoperative mortality and morbidity. Patients classified as very frail have 30-day and 180-day mortality rates of approximately 10% and 40%, respectively, even following minor surgeries.

A new tool for assessing frailty, the 5-item modified frailty index (mFI-5), has recently been developed using data from the National Surgical Quality Improvement Program (NSQIP) database. This simplified scale, which consists of only five items, has demonstrated superior predictive ability compared to previously utilized tools. The mFI-5 has been studied across various surgical populations and has been found to be associated with unfavorable postoperative outcomes. However, there are limited studies examining its utility in urologic surgery, and no reports has investigated the association between frailty and minimally invasive urologic procedures. Therefore, the present study aimed to investigate the correlation between the modified 5-item frailty index and postoperative mortality and complications among frail patients who undergo urologic surgery.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients who underwent urologic procedures were recruited

(Included procedures : all urologic oncology surgeries, suburethral sling placement and laparoscopic pyeloplasty, transurethral resection of the prostate, transurethral resection of the bladder tumor, ureteroscopy, hydrocelectomy, orchiectomy, spermatocelectomy, epididymectomy, and varicocelectomy.)

Exclusion Criteria:

* Incomplete information of baseline parameters

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Surgical cases from 2015 to 2020 NSQIP dataset
Sampling Method: Non-Probability Sample
Enrollment: 317076 (Actual)
Dates: Start 2023-01-01 (Actual); Primary Completion 2023-03-16 (Actual); Study Completion 2023-05-15 (Actual)

PRIMARY OUTCOMES:
postoperative mortality | within 30 days after the primary procedure
  postoperative in-hospital mortality

SECONDARY OUTCOMES:
postoperative complications | within 30 days after the primary procedure
  cardiovascular events, cerebrovascular events, pneumonia, surgical site infection, sepsis, bleeding, mechanical ventilation >48 hrs, reoperation, readmission, and length of hospital stay.

CONTACTS AND LOCATIONS:
Overall Officials: Chao-Shun Lin, PhD, Study Chair — Department of Anesthesiology, Taipei Medical University Hospital, 252 Wuxing St., Taipei 110 Taiwan
Locations (1):
- Taipei Medical University Hospital, Taipei, Taiwan